CLINICAL TRIAL: NCT01310413
Title: Safety and Immunogenicity of Monovalent H5N1 Vaccine GSK1557484A in Children 6 Months to < 18 Years of Age
Brief Title: Monovalent H5N1 Vaccine GSK1557484A in Children 6 Months to < 18 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114464; 2012-001683-29 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-03-08 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Influenza; Influenza Vaccines
Keywords: Influenza; H5N1; Pandemic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (7):
- Influenza A (H5N1) adjuvanted 6-<36M Group (Experimental): Subjects aged at enrolment between 3 and 36 months, 36 months excluded, received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine
- Influenza A (H5N1) Virus monovalent vaccine 3-<9Y Group (Experimental): Subjects aged at enrolment between 3 and 9 years, 9 years excluded, received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine
- Influenza A (H5N1) Virus monovalent vaccine 9-<18Y Group (Experimental): Subjects aged at enrolment between 9 and 18 years, 18 years excluded, received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine
- Placebo 6-<36M Group (Placebo Comparator): Subjects aged at enrolment between 3 and 36 months, 36 months excluded, received 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: Saline placebo
- Placebo 3-<9Y Group (Placebo Comparator): Subjects aged at enrolment between 3 and 9 years, 9 years excluded, received 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: Saline placebo
- Placebo 9-<18Y Group (Placebo Comparator): Subjects aged at enrolment between 9 and 18 years, 18 years excluded, received 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: Saline placebo
- Placebo/Influenza A (H5N1) adjuvanted Group (Experimental): Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6-<36M, Placebo 3-<9Y or Placebo 9-<18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 of was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus monovalent vaccine — All subjects will receive 2 doses administered as an intramuscular (IM) injection.
  Arms: Influenza A (H5N1) Virus monovalent vaccine 3-<9Y Group; Influenza A (H5N1) Virus monovalent vaccine 9-<18Y Group; Influenza A (H5N1) adjuvanted 6-<36M Group; Placebo/Influenza A (H5N1) adjuvanted Group
Biological: Saline placebo — All subjects will receive 2 doses administered as an intramuscular (IM) injection.
  Arms: Placebo 3-<9Y Group; Placebo 6-<36M Group; Placebo 9-<18Y Group

SUMMARY:
This study will assess safety and immunogenicity of GSK Biologicals' H5N1 flu candidate vaccine GSK1557484A in children 6 months to < 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female child >= 6 months and < 18 years of age at the time of first vaccination.
* Written informed consent obtained from the subject's parent/guardian.
* Documentation of assent for children 9 to < 18 years of age (or as deemed mandatory by local practice).
* Satisfactory baseline medical assessment by history and physical examination
* Parent/guardian and subject access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Parents/guardians and subjects who the investigator believes understand the requirements of the protocol and can and will comply with them.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential must

  * have practiced adequate contraception for 30 days prior to vaccination, and
  * have a negative pregnancy test on the day of each vaccination, and
  * have agreed to continue adequate contraception for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an H5N1 virus.
* Previous vaccination at any time with an H5N1 vaccine.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine/product, or planned use during the study period.
* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Presence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject or parent/guardian unable/unlikely to provide accurate safety reports.
* Evidence of current subject or parent/guardian substance abuse, including alcohol, by medical history.
* Presence of a temperature >= 38.0ºC by any method, or acute symptoms greater than "mild" severity on the scheduled date of first dose.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Receipt of systemic glucocorticoids within 1 month prior to first dose of test article or any other cytotoxic or immunosuppressive drug within 6 months prior to first dose of test article. Receipt of any immunoglobulins and/or any blood products within 3 months of first test article administration or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Administration of an inactivated seasonal influenza vaccine within 14 days, or of a live, attenuated seasonal influenza vaccine within 30 days before the first test article dose, or of any other vaccine(s) not foreseen by the study protocol within 30 days before the first test article dose.
* Planned administration of any vaccine(s) not foreseen by the study protocol through completion of the "Day 42" visit.
* Any known or suspected allergy to any constituent of influenza vaccines or history of severe reaction to any previous influenza vaccination.
* Known pregnancy, or a positive urine pregnancy test result prior to each test article dose.
* Lactating or nursing.
* Child in care.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 842 (Actual)
Dates: Start 2011-03-07 (Actual); Primary Completion 2011-07-21 (Actual); Study Completion 2014-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (11):
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Angelo, Texas
- Canada (4):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Izurieta P et al. (2018) Reactogenicity and safety of AS03B-adjuvanted H5N1 influenza vaccine in children: an open-label, one-way, crossover trial. Asian Biomed (Res Rev News). 11(4):359-364.
- [Background] Kosalaraksa P, Jeanfreau R, Frenette L, Drame M, Madariaga M, Innis BL, Godeaux O, Izurieta P, Vaughn DW. AS03B-adjuvanted H5N1 influenza vaccine in children 6 months through 17 years of age: a phase 2/3 randomized, placebo-controlled, observer-blinded trial. J Infect Dis. 2015 Mar 1;211(5):801-10. doi: 10.1093/infdis/jiu548. Epub 2014 Oct 6. PMID 25293368
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114464 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included a first 385-days Blinded Phase (all subjects), followed by a 385-days Unblinded Phase. In this phase, subjects who received the placebo in the Blinded Phase were offered, after completing the Blinded Phase, 2 doses of Influenza A (H5N1) Virus monovalent vaccine administered for Dose 1 within a short delay of Day 385 (Day U0).
Pre-assignment Details: A total of 842 subjects were enrolled in the study in its Blinded Phase part. This number was later amended down to 838, following corrections for wrong subject number allocation and randomization errors.
Groups:
- Influenza A (H5N1) Adjuvanted 3-<9Y Group: Subjects aged at enrolment between 3 and 9 years, 9 years excluded, received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
- Influenza A (H5N1) Adjuvanted 9-<18Y Group: Subjects aged at enrolment between 9 and 18 years, 18 years excluded, received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
- Placebo 6-<36M Group: Subjects aged at enrolment between 3 and 36 months, 36 months excluded, received 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly. For children aged up to 12 months, 12 months excluded (<12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
- Placebo/Influenza A (H5N1) Adjuvanted Group: Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6-<36M, Placebo 3-<9Y or Placebo 9-<18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
Period: Day 0 to Day 385
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group | Placebo/Influenza A (H5N1) Adjuvanted Group
Started | 199 | 198 | 210 | 75 | 76 | 80 | 0 (This group is only followed during the Unblinded Phase of the study, from Days U0 to U385.)
Completed | 172 | 190 | 203 | 67 | 73 | 77 | 0 (This group is only followed during the Unblinded Phase of the study, from Days U0 to U385.)
Not Completed | 27 | 8 | 7 | 8 | 3 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 2 | 0 | 2 | 1 | 1 | 0
Not completed — Lost to Follow-up | 18 | 3 | 3 | 5 | 1 | 2 | 0
Not completed — Migrated/moved from study area | 3 | 3 | 1 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 3 | 0 | 0 | 0 | 0
Period: From Day U0 to Day U385
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group | Placebo/Influenza A (H5N1) Adjuvanted Group
Started | 0 (Subjects from this group were not included in Day U0 to Day U42 analysis as per study protocol.) | 0 (Subjects from this group were not included in Day U0 to Day U42 analysis as per study protocol.) | 0 (Subjects from this group were not included in Day U0 to Day U42 analysis as per study protocol.) | 0 (Eligible subjects who provided consent were included in Placebo/Influenza A (H5N1) Adjuvanted Group.) | 0 (Eligible subjects who provided consent were included in Placebo/Influenza A (H5N1) Adjuvanted Group.) | 0 (Eligible subjects who provided consent were included in Placebo/Influenza A (H5N1) Adjuvanted Group.) | 155 (Upto Day U42)
Completed | 0 (Subjects from this group were not included in Day U0 to Day U42 analysis as per study protocol.) | 0 (Subjects from this group were not included in Day U0 to Day U42 analysis as per study protocol.) | 0 (Subjects from this group were not included in Day U0 to Day U42 analysis as per study protocol.) | 0 (Eligible subjects who provided consent were included in Placebo/Influenza A (H5N1) Adjuvanted Group.) | 0 (Eligible subjects who provided consent were included in Placebo/Influenza A (H5N1) Adjuvanted Group.) | 0 (Eligible subjects who provided consent were included in Placebo/Influenza A (H5N1) Adjuvanted Group.) | 152 (Upto Day U42)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group | Total
Number analyzed (Participants) | 199 | 198 | 210 | 75 | 76 | 80 | 838
Age, Continuous [Mean (Standard Deviation); unit: Months] | 21.7 (8.17) | 70.5 (21.71) | 160.8 (28.21) | 22.6 (8.17) | 65.2 (20.2) | 156.0 (31.29) | 84.9 (61.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 90 | 103 | 39 | 35 | 42 | 401
  Male | 107 | 108 | 107 | 36 | 41 | 38 | 437

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroprotected for Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: A seroprotected subject against the a/Indonesia/5/2005 (A/INDO) virus strain was defined as a subject with H5N1 reciprocal haemagglutination inhibition (HI) antibody titers greater than or equal to (>=) the seroprotection cut-off of 1:40.
Time Frame: At Day 42.
Population: The analyses were performed on According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects who received 2 doses of the study vaccine/placebo at Days 0 and 21 and for whom assay results for antibodies against vaccine-homologous H5N1 HA antigen for the blood samples taken at Days 0 and 42 were available.
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 175 | 185 | 203 | 64 | 71 | 76
Subject | 175 | 184 | 201 | 0 | 0 | 1

2. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: HI antibody titers against the H5N1 A/Indonesia virus strain (A/INDO) were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of higher than or equal to (>=) 1:10.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 182 | 184 | 204 | 67 | 71 | 76
Titer
  A/INDO, Day 0 [N=182;184;204;67;71;76] | 5.3 [5.1 to 5.5] | 5.6 [5.3 to 5.9] | 5.7 [5.4 to 6.1] | 5.3 [5.0 to 5.7] | 5.6 [5.1 to 6.0] | 5.4 [5.1 to 5.8]
  A/INDO, Day 21 [N=179;184;204;67;70;76] | 38.7 [33.9 to 44.2] | 44.6 [39.2 to 50.9] | 35.3 [31.7 to 39.5] | 5.2 [5.0 to 5.4] | 5.4 [5.0 to 5.7] | 5.4 [5.1 to 5.7]

3. Secondary Outcome: Number of Subjects Seroprotected for Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: as for outcome 1
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 182 | 184 | 204 | 67 | 71 | 76
Subject
  A/INDO, Day 0 [N=182;184;204;67;71;76] | 1 | 2 | 1 | 0 | 0 | 0
  A/INDO, Day 21 [N=179;184;204;67;70;76] | 105 | 110 | 108 | 0 | 1 | 0

4. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Description: A subject seroconverted for HI antibodies against the H5N1 A/Indonesia virus strain (A/INDO) was defined as a vaccinee with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer higher than or equal to (>=) 1:40, or with a pre-vaccination titer >= 1:10 and at least a 4-fold increase in post-vaccination titer.
  As the analyses were performed and disclosed stepwise - i.e. as soon as a study phase was completed - several releases of the CTRS (result summaries) were published. To generate an integrated Clinical Study Report, one set of domain datasets covering all analyses was used and the Adapted ATP cohort for immunogenicity has been defined. As a consequence, some of the data previously disclosed and based on ATP cohort for immunogenicity at Day 42, Day 182 and Day 385 have been replaced in this summary with data generated with the Adapted ATP cohort for immunogenicity.
Time Frame: At Days 21 and 42
Population: Adapted ATP cohort for immunogenicity included all evaluable subjects for which Day 21 and Day 42 data were obtained from the ATP cohort for immunogenicity at Day 42; Day 182 data were obtained from the ATP cohort for immunogenicity at Day 182, and Day 385 data were obtained from the ATP cohort for immunogenicity at Day 385.
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 179 | 185 | 204 | 67 | 71 | 76
Subject
  A/INDO, Day 21 [N=179;183;204;67;70;76] | 103 | 107 | 105 | 0 | 0 | 0
  A/INDO, Day 42 [N=175;184;203;64;71;76] | 175 | 183 | 201 | 0 | 0 | 1

5. Secondary Outcome: Geometric Mean Increase (GMI) for Haemagglutination Inhibition (HI) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Description: GMI also known as the seroconversion factor (SCF) or geometric mean fold rise (GMFR) was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titre to the pre-vaccination reciprocal HI titre for the vaccine virus.
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 179 | 185 | 204 | 67 | 71 | 76
Ratio
  A/INDO, Day 21 [N=179;183;204;67;70;76] | 7.3 [6.4 to 8.4] | 8.0 [7.0 to 9.1] | 6.2 [5.5 to 6.9] | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.1]
  A/INDO, Day 42 [N=175;184;203;64;71;76] | 148.5 [134.5 to 164.1] | 96.9 [85.3 to 110.1] | 72.4 [63.9 to 82.0] | 1.0 [0.9 to 1.0] | 1.0 [0.9 to 1.0] | 1.1 [1.0 to 1.2]

6. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: HI antibody titers against the H5N1 A/Indonesia virus strain (A/INDO) were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of higher than or equal to (>=) 1:10.
  Adapted ATP cohort for immunogenicity included all evaluable subjects for which Day 21 and Day 42 data were obtained from the ATP cohort for immunogenicity at Day 42; Day 182 data were obtained from the ATP cohort for immunogenicity at Day 182, and Day 385 data were obtained from the ATP cohort for immunogenicity at Day 385.
Time Frame: At Day 0 and Day 182.
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titre
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 107 | 101 | 100 | 36 | 37 | 35
Titre
  A/INDO, Day 0 [N=107;101;100;36;37;35] | 5.1 [5.0 to 5.2] | 5.2 [5.0 to 5.4] | 5.6 [5.2 to 6.0] | 5.3 [4.9 to 5.7] | 5.2 [4.8 to 5.8] | 5.4 [4.8 to 6.0]
  A/INDO, Day 182 [N=84;89;87;29;34;31] | 90.6 [78.1 to 105.0] | 57.4 [50.8 to 64.9] | 50.2 [43.3 to 58.2] | 5.0 [5.0 to 5.0] | 5.4 [4.9 to 6.0] | 5.4 [4.9 to 5.9]

7. Secondary Outcome: Number of Subjects Seroprotected as Regards Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: A seroprotected subject against the a/Indonesia/5/2005 (A/INDO) virus strain was defined as a subject with H5N1 reciprocal haemagglutination inhibition (HI) antibody titers greater than or equal to (>=) the seroprotection cut-off of 1:40.
  As the analyses were performed and disclosed stepwise - i.e. as soon as a study phase was completed - several releases of the CTRS (result summaries) were published. To generate an integrated Clinical Study Report, one set of domain datasets covering all analyses was used and the Adapted ATP cohort for immunogenicity has been defined. As a consequence, some of the data previously disclosed and based on ATP cohort for immunogenicity at Day 42, Day 182 and Day 385 have been replaced in this summary with data generated with the Adapted ATP cohort for immunogenicity.
Time Frame: At Day 0 and Day 182
Population: as for outcome 4
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 182 | 184 | 204 | 67 | 71 | 76
Subject
  A/INDO, Day 0 [N=182;184;204;67;71;76] | 1 | 2 | 1 | 0 | 0 | 0
  A/INDO, Day 182 [N=84;89;87;29;34;31] | 80 | 75 | 63 | 0 | 0 | 0

8. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain
Description: HI antibody titers against the H5N1 A/Indonesia virus strain (A/INDO) were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of higher than or equal to (>=) 1:10.
  As the analyses were performed and disclosed stepwise - i.e. as soon as a study phase was completed - several releases of the CTRS (result summaries) were published. To generate an integrated Clinical Study Report, one set of domain datasets covering all analyses was used and the Adapted ATP cohort for immunogenicity has been defined. As a consequence, some of the data previously disclosed and based on ATP cohort for immunogenicity at Day 42, Day 182 and Day 385 have been replaced in this summary with data generated with the Adapted ATP cohort for immunogenicity.
Time Frame: At Day 42.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 175 | 185 | 203 | 64 | 71 | 76
Titer | 777.1 [705.6 to 855.9] | 543.8 [484.9 to 609.8] | 416.2 [371.5 to 466.2] | 5.1 [4.9 to 5.3] | 5.4 [5.0 to 5.7] | 5.8 [5.3 to 6.3]

9. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Description: A subject seroconverted for HI antibodies against the H5N1 A/Indonesia virus strain (A/INDO) was defined as a vaccinee with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer higher than or equal to (>=) 1:40, or with a pre-vaccination titer >= 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 182
Population: The analyses were performed on According-to-Protocol (ATP) cohort for immunogenicity at Day 182, which included 50% of evaluable subjects who received 2 doses of the study vaccine/placebo at Days 0 and 21 and for whom assay results for antibodies against vaccine-homologous H5N1 HA antigen for the blood samples taken at Days 0 and 182 were available
Measure: Number; unit: Subject
Groups:
- Influenza A (H5N1) Adjuvanted 3-<9Y Group: SSubjects aged at enrolment between 3 and 9 years, 9 years excluded, received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly, Dose 1 in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 84 | 89 | 87 | 29 | 34 | 31
Subject | 80 | 75 | 61 | 0 | 0 | 0

10. Secondary Outcome: Geometric Mean Increase (GMI) for Haemagglutination Inhibition (HI) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Description: as for outcome 5
Time Frame: At Day 182
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 84 | 89 | 87 | 29 | 34 | 31
Ratio | 17.8 [15.3 to 20.8] | 11.0 [9.7 to 12.4] | 8.8 [7.5 to 10.4] | 1.0 [0.9 to 1.0] | 1.1 [1.0 to 1.2] | 1.0 [0.9 to 1.2]

11. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: as for outcome 8
Time Frame: At Day 0 and Day 385
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 182 | 184 | 204 | 67 | 71 | 76
Titer
  A/INDO, Day 0 [N=182;184;204;67;71;76] | 5.3 [5.1 to 5.5] | 5.6 [5.3 to 5.9] | 5.7 [5.4 to 6.1] | 5.3 [5.0 to 5.7] | 5.6 [5.1 to 6.0] | 5.4 [5.1 to 5.8]
  A/INDO, Day 385 [N=63;85;95;26;34;36] | 65.6 [55.9 to 76.9] | 32.8 [28.1 to 38.4] | 21.6 [18.6 to 25.1] | 5.1 [4.9 to 5.4] | 5.4 [4.9 to 5.8] | 5.3 [4.8 to 5.9]

12. Secondary Outcome: Number of Subjects Seroprotected for Haemagglutination Inhibition (HI) Antibody Titers Against the H5N1 A/Indonesia Virus Strain.
Description: as for outcome 7
Time Frame: At Day 0 and Day 385
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 182 | 184 | 204 | 67 | 71 | 76
Subjects
  A/INDO, Day 0 [N=182, 184,204,67,71,76] | 1 | 2 | 1 | 0 | 0 | 0
  A/INDO, Day 385 [N=63;85;95;26;34;36] | 54 | 47 | 27 | 0 | 0 | 0

13. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Description: as for outcome 9
Time Frame: At Day 385
Population: The analyses were performed on According-to-Protocol (ATP) cohort for immunogenicity at Day 385, which included 50% of evaluable subjects who received 2 doses of the study vaccine/placebo at Days 0 and 21 and for whom assay results for antibodies against vaccine-homologous H5N1 HA antigen for the blood samples taken at Days 0 and 385 were available
Measure: Number; unit: Subjects
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 63 | 85 | 95 | 26 | 34 | 36
Subjects | 53 | 45 | 23 | 0 | 0 | 0

14. Secondary Outcome: Geometric Mean Increase (GMI) for Haemagglutination Inhibition (HI) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Description: GMI also known as the seroconversion factor (SCF) or geometric mean fold rise (GMFR) was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination reciprocal HI titer for the vaccine virus.
Time Frame: At Day 385.
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 63 | 85 | 95 | 26 | 34 | 36
Fold increase | 12.1 [10.3 to 14.2] | 5.5 [4.7 to 6.6] | 3.6 [3.1 to 4.3] | 1.0 [0.9 to 1.1] | 0.9 [0.8 to 1.0] | 1.0 [0.8 to 1.1]

15. Secondary Outcome: Microneutralization (MN) Antibody Titers Against the H5N1 A/Indonesia and H5N1 A/Vietnam Virus Strains.
Description: MN HI antibody titers against the H5N1 A/Indonesia (A/INDO) and H5N1 A/Vietnam (A/VIET) virus strains were expressed as geometric mean titers (GMTs). The cut-off of the assay was the seropositivity cut-off of higher than or equal to (>=) 1:28.
Time Frame: At Days 0, 42, 182 and 385
Population: Analysis was done on the Day 42, 182 and 385 ATP cohorts for immunogenicity, that is, 50 percent of the evaluable subjects with 2 doses of vaccine/placebo administered and for whom assay results for antibodies against vaccine-homologous H5N1 haemagglutinin (HA) antigen were available for the Days 0, 42, 182 and 385 time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 36 | 39 | 40 | 10 | 11 | 11
Titer
  A/INDO, Day 0 [N=36;37;40;7;10;11] | 14.00 [14.00 to 14.00] | 15.67 [14.37 to 17.08] | 15.54 [14.13 to 17.09] | 15.46 [12.13 to 19.70] | 14.00 [14.00 to 14.00] | 14.91 [12.96 to 17.16]
  A/INDO, Day 42 [N=34;37;40;6;10;11] | 855.62 [597.88 to 1224.47] | 657.60 [453.13 to 954.33] | 380.62 [277.43 to 522.20] | 14.00 [14.00 to 14.00] | 14.00 [14.00 to 14.00] | 14.91 [12.96 to 17.16]
  A/INDO, Day 182 [N=33;39;33;10;10;9] | 216.82 [162.03 to 290.14] | 130.32 [107.30 to 158.26] | 104.18 [86.95 to 124.82] | 16.11 [11.73 to 22.13] | 14.00 [14.00 to 14.00] | 17.67 [12.08 to 25.86]
  A/INDO, Day 385 [N=25;33;37;8;11;9] | 166.64 [135.90 to 204.32] | 108.59 [87.88 to 134.19] | 82.26 [67.27 to 100.59] | 15.27 [12.44 to 18.74] | 14.91 [12.96 to 17.16] | 16.33 [12.91 to 20.66]
  A/VIET, Day 0 [N=36;36;40;7;10;11] | 14.83 [13.89 to 15.84] | 19.84 [16.82 to 23.40] | 24.88 [20.75 to 29.85] | 17.11 [10.47 to 27.95] | 16.08 [13.05 to 19.82] | 20.47 [14.82 to 28.26]
  A/VIET, Day 42 [N=34;37;40;6;10;11] | 68.18 [58.05 to 80.07] | 71.15 [61.62 to 82.15] | 65.25 [57.03 to 74.64] | 17.69 [9.69 to 32.28] | 19.87 [12.97 to 30.43] | 28.14 [19.53 to 40.54]
  A/VIET, Day 182 [N=33;39;33;10;10;9] | 48.77 [36.56 to 65.06] | 44.11 [36.19 to 53.77] | 61.67 [51.38 to 74.01] | 19.82 [12.22 to 32.14] | 17.24 [13.56 to 21.90] | 24.14 [14.29 to 40.78]
  A/VIET, Day 385 [N=25;33;37;8;11;9] | 59.83 [48.09 to 74.43] | 38.62 [30.60 to 48.73] | 47.73 [38.76 to 58.79] | 14.00 [14.00 to 14.00] | 18.07 [12.34 to 26.47] | 35.42 [19.45 to 64.49]

16. Secondary Outcome: Number of Subjects Seropositive for Microneutralization (MN) Antibodies Against the H5N1 A/Indonesia Virus Strain.
Time Frame: At Days 0 and 42
Population: Analysis was done on the Day 42 According-to-Protocol cohort for immunogenicity, that is, all evaluable subjects with 2 doses of vaccine/placebo administered and for whom assay results for antibodies against vaccine-homologous H5N1 haemagglutinin (HA) antigen were available for the Days 0 and 42 time points.
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Virus Monovalent Vaccine 3-<9Y Group | Influenza A (H5N1) Virus Monovalent Vaccine 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 36 | 37 | 40 | 7 | 10 | 11
Subject
  At Day 0 | 0 | 6 | 5 | 1 | 0 | 1
  At Day 42 | 34 | 37 | 40 | 0 | 0 | 1

17. Secondary Outcome: Vaccine Response Rate (VRR) for Microneutralization (MN) Antibodies Against the H5N1 A/Indonesia and H5N1 A/Vietnam Virus Strains.
Description: VRR for MN was defined as as the incidence rate of vaccinees with a 4-fold increase in post vaccination reciprocal titer relative to Day 0.
Time Frame: At Day 42
Population: as for outcome 16
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted 6-<36M Group | Influenza A (H5N1) Adjuvanted 3-<9Y Group | Influenza A (H5N1) Adjuvanted 9-<18Y Group | Placebo 6-<36M Group | Placebo 3-<9Y Group | Placebo 9-<18Y Group
Number analyzed (Participants) | 34 | 37 | 40 | 6 | 11 | 11
Subject
  A/INDO [N=34;37;40;6;10;11] | 34 | 37 | 39 | 0 | 0 | 0
  A/VIET [N=34;36;40;6;10;11] | 30 | 26 | 16 | 0 | 1 | 0

18. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. "Any" was defined as any occurrence of the specified solicited local symptom reported, regardless of intensity. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 100 millimeter (mm).
Time Frame: During the 7-day (Days 0-6) post-vaccination periods post Doses 1 and 2 of vaccine/placebo, across doses (Year 1)
Population: Analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented, solely on subjects with results available/accessible.
Measure: Number; unit: Subject
Groups:
- Influenza A (H5N1) Adjuvanted Group: This group results from the pooling of the Influenza A (H5N1) adjuvanted 6-<36M, Influenza A (H5N1) adjuvanted 3-<9Y and Influenza A (H5N1) adjuvanted months and 18 years, 18 years excluded, who received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
- Placebo Group: This group results from the pooling of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 603 | 229
Subject
  Any pain | 405 | 69
  Grade 3 pain | 25 | 4
  Any redness | 29 | 0
  Grade 3 redness | 1 | 0
  Any swelling | 41 | 1
  Grade 3 swelling | 1 | 0

19. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain and swelling. "Any" was defined as any occurrence of the specified solicited local symptom reported, regardless of intensity. Grade 3 pain was defined as pain that prevented normal activity. Grade 3 redness and swelling were defined as redness/swelling above 100 millimeter (mm).
Time Frame: During the 7-day (Days U0-U6) post-vaccination periods post Doses 1 and 2 of vaccine/placebo, across doses (Year 2)
Population: Analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Number; unit: Subject
Groups:
- Placebo/Placebo/ Influenza A (H5N1) Adjuvanted Group: Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6-<36M, Placebo 3-<9Y or Placebo 9-<18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
Arm/Group | Placebo/Placebo/ Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 154
Subject
  Any Pain | 111
  Grade 3 Pain | 8
  Any Redness | 6
  Grade 3 Redness | 0
  Any Swelling | 5
  Grade 3 Swelling | 0

20. Secondary Outcome: Number of Subjects of Less Than 6 Years of Age Reporting Solicited General Symptoms.
Description: Solicited general symptoms assessed in subjects of less than 6 years of age were drowsiness, irritability/fussiness, loss of appetite and fever [axillary temperature (T) higher than or equal to (>=) 38.0 degrees Celsius (°C)]. "Any" was defined as any occurrence of the specified solicited general symptom reported, regardless of intensity or relationship to vaccination. Grade 3 was defined as a general symptom that prevented normal activity. Related was defined as a general symptom assessed by the investigator as causally related to the study vaccination. Any fever was defined as axillary temperature above 38.0 degrees Celsius (°C). Grade 3 fever was axillary temperature >= 39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination periods post Doses 1 and 2 of vaccine/placebo, across doses (Year 1)
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Influenza A (H5N1) Adjuvanted Group: This group results from the pooling of the Influenza A (H5N1) adjuvanted 6-<36M, PInfluenza A (H5N1) adjuvanted 3-<9Y and Influenza A (H5N1) adjuvanted 9-<18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 294 | 122
Subject
  Any Drowsiness | 101 | 29
  Grade 3 Drowsiness | 9 | 2
  Related Drowsiness | 81 | 21
  Any Irritability/fussiness | 128 | 40
  Grade 3 Irritability/fussiness | 10 | 2
  Related Irritability/fussiness | 111 | 33
  Any Loss of appetite | 79 | 29
  Grade 3 Loss of appetite | 8 | 4
  Related Loss of appetite | 63 | 20
  Any Fever | 59 | 21
  Grade 3 Fever | 14 | 5
  Related Fever | 41 | 14

21. Secondary Outcome: Number of Subjects of Less Than 6 Years of Age Reporting Solicited General Symptoms.
Description: Solicited general symptoms assessed in subjects of less than 6 years of age were drowsiness, irritability/fussiness, loss of appetite and fever [axillary temperature (T) higher than or equal to (>=) 38.0 degrees Celsius (°C)]. "Any" was defined as any occurrence of the specified solicited general symptom reported, regardless of intensity or relationship to vaccination. Grade 3 was defined as a general symptom that prevented normal activity. Related was defined as a general symptom assessed by the investigator as causally related to the study vaccination. Any fever was defined as axillary temperature above 38.0 degrees Celsius (°C). Grade 3 fever was axillary temperature >=39.0°C.
Time Frame: During the 7-day (Days U0-U6) post-vaccination periods post Doses 1 and 2 of vaccine/placebo, across doses (Year 2)
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Placebo/ Influenza A (H5N1) Adjuvanted Group: Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6-<36M, Placebo 3-<9Y or Placebo 9-<18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
Arm/Group | Placebo/ Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 79
Subject
  Any Drowsiness | 23
  Grade 3 Drowsiness | 1
  Related Drowsiness | 17
  Any Irritability/Fussiness | 28
  Grade 3 Irritability/Fussiness | 1
  Related Irritability/Fussiness | 23
  Any Loss of appetite | 18
  Grade 3 Loss of appetite | 0
  Related Loss of appetite | 13
  Any Fever | 4
  Grade 3 Fever | 2
  Related Fever | 3

22. Secondary Outcome: Number of Subjects at Least 6 Years of Age Reporting Solicited General Symptoms.
Description: Solicited general symptoms assessed in subjects of at least 6 years of age were fatigue, gastrointestinal symptoms, headache, joint pain at other location, muscle aches, shivering, sweating and fever [axillary temperature (T) >= 38.0 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diaorrhea and/or abdominal pain. "Any" was defined as any occurrence of the specified solicited general symptom reported, regardless of intensity or relationship to vaccination. Grade 3 was defined as a general symptom that prevented normal activity. Related was defined as a general symptom assessed by the investigator as causally related to the study vaccination. Grade 3 fever was axillary temperature >= 39.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination periods post Doses 1 and 2 of vaccine/placebo, across doses (Year 1)
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Influenza A (H5N1) Adjuvanted Group: This group results from the pooling of the Influenza A (H5N1) adjuvanted 6-<36M, Influenza A (H5N1) adjuvanted 3-<9Y and Influenza A (H5N1) adjuvanted 9-<18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 309 | 107
Subject
  Any fatigue | 89 | 19
  Grade 3 fatigue | 4 | 2
  Related fatigue | 77 | 16
  Any gastrointestinal symptoms | 43 | 18
  Grade 3 gastrointestinal symptoms | 4 | 2
  Related gastrointestinal symptoms | 27 | 11
  Any headache | 100 | 18
  Grade 3 headache | 8 | 3
  Related headache | 87 | 15
  Any joint pain | 50 | 9
  Grade 3 joint pain | 2 | 0
  Related joint pain | 43 | 8
  Any muscle aches | 123 | 17
  Grade 3 muscle aches | 7 | 1
  Related muscle aches | 114 | 14
  Any shivering | 25 | 7
  Grade 3 shivering | 2 | 1
  Related shivering | 19 | 5
  Any sweating | 25 | 4
  Grade 3 sweating | 2 | 0
  Related sweating | 22 | 1
  Any fever | 19 | 3
  Grade 3 fever | 5 | 1
  Related fever | 13 | 2

23. Secondary Outcome: Number of Subjects at Least 6 Years of Age Reporting Solicited General Symptoms.
Description: as for outcome 22
Time Frame: During the 7-day (Days U0-U6) post-vaccination periods post Doses 1 and 2 of vaccine/placebo, across doses (Year 2)
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Placebo/Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 75
Subject
  Any Fatigue | 18
  Grade 3 Fatigue | 1
  Related Fatigue | 13
  Any Gastrointestinal | 7
  Grade 3 Gastrointestinal | 0
  Related Gastrointestinal | 5
  Any Headache | 24
  Grade 3 Headache | 1
  Related Headache | 20
  Any Increased Sweating | 5
  Grade 3 Increased Sweating | 0
  Related Increased Sweating | 3
  Any Joint Pain | 14
  Grade 3 Joint Pain | 0
  Related Joint Pain | 12
  Any Muscle Aches | 34
  Grade 3 Muscle Aches | 0
  Related Muscle Aches | 28
  Any Shivering (Chills) | 7
  Grade 3 Shivering (Chills) | 2
  Related Shivering (Chills) | 4
  Any Fever | 1
  Grade 3 Fever | 0
  Related Fever | 0

24. Secondary Outcome: Number of Subjects With Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination. Any MAE was defined as atleast 1 MAE experienced.
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject | 189 | 77

25. Secondary Outcome: Number of Subjects With Medically-attended Adverse Events (MAEs)
Description: as for outcome 24
Time Frame: From Day U0 up to Day U385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Placebo/ Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 155
Subject | 36

26. Secondary Outcome: Number of Subjects With Any Potential Immune-Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) were defined as a subset of adverse events that included both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which might or might not have an autoimmune aetiology. "Any pIMD" was defined as at least one pIMD experienced by the study subject.
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Influenza A (H5N1) Adjuvanted Group: This group results from the pooling of the PInfluenza A (H5N1) adjuvanted 6-<36M, Influenza A (H5N1) adjuvanted 3-<9Y and Influenza A (H5N1) adjuvanted 9-<18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject | 1 | 1

27. Secondary Outcome: Number of Subjects With Any Potential Immune-Mediated Diseases (pIMDs)
Description: as for outcome 26
Time Frame: From Day U0 to Day U385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Placebo/ Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 155
Subject | 0

28. Secondary Outcome: Number of Subjects Reporting Pregnancies, and Outcomes of These Reported Pregnancies
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  Subject(s) with any pregnancy | 2 | 0
  Subject(s) with related pregnancy | 0 | 0
  Spontaneous abortion | 1 | 0
  Healthy live birth | 1 | 0

29. Secondary Outcome: Number of Subjects Reporting Pregnancies, and Outcomes of These Reported Pregnancies
Time Frame: From Day U0 to Day U385
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Placebo/ Influenza A (H5N1) Adjuvanted Group: Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6-<36M, Placebo 3-<9Y or Placebo 9-<18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 of was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
Arm/Group | Placebo/ Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 155
Subject | 0

30. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Alanine Aminotransferase (ALAT) and Aspartate Aminotransferase (ASAT)
Description: Subjects were categorized according to their results at pre-vaccination (PRE), Day 42, Day 182 and Day 385 which were normal, above normal, below the normal ranges or unknown.
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Placebo Group: This group results from the pooling of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly. For children aged up to 12 months, 12 months excluded (<12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 606 | 231
Subject
  ALAT, PRE Unknown [N=606,231] | 15 | 4
  ALAT, PRE Below [N=606,231] | 0 | 0
  ALAT, PRE Normal [N=606,231] | 586 | 221
  ALAT, PRE Above [N=606,231] | 5 | 6
  ALAT, Day 42 Unknown [N=583,220] | 17 | 4
  ALAT, Day 42 Below [N=583,220] | 0 | 0
  ALAT, Day 42 Normal [N=583,220] | 562 | 212
  ALAT, Day 42 Above [N=583,220] | 4 | 4
  ALAT, Day 182 Unknown [N=304,110] | 6 | 0
  ALAT, Day 182 Below [N=304,110] | 0 | 0
  ALAT, Day 182 Normal [N=304,110] | 289 | 110
  ALAT, Day 182 Above [N=304,110] | 9 | 0
  ALAT, Day 385 Unknown [N=251,104] | 5 | 0
  ALAT, Day 385 Below [N=251,104] | 0 | 0
  ALAT, Day 385 Normal [N=251,104] | 245 | 100
  ALAT, Day 385 Above [N=251,104] | 1 | 4
  ASAT, PRE Unknown [N=606,231] | 15 | 4
  ASAT, PRE Below [N=606,231] | 0 | 0
  ASAT, PRE Normal [N=606,231] | 577 | 219
  ASAT, PRE Above [N=606,231] | 14 | 8
  ASAT, Day 42 Unknown [N=583,220] | 19 | 4
  ASAT, Day 42 Below [N=583,220] | 0 | 0
  ASAT, Day 42 Normal [N=583,220] | 552 | 208
  ASAT, Day 42 Above [N=583,220] | 12 | 8
  ASAT, Day 182 Unknown [N=304,110] | 8 | 0
  ASAT, Day 182 Below [N=304,110] | 0 | 0
  ASAT, Day 182 Normal [N=304,110] | 284 | 108
  ASAT, Day 182 Above [N=304,110] | 12 | 2
  ASAT, Day 385 Unknown [N=251,104] | 7 | 0
  ASAT, Day 385 Below [N=251,104] | 0 | 0
  ASAT, Day 385 Normal [N=251,104] | 240 | 100
  ASAT, Day 385 Above [N=251,104] | 4 | 4

31. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Total Bilirubin (T-BIL) and Bilirubin Conjugated/Direct (BIL-C/D)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 606 | 231
Subject
  T-BIL, PRE Unknown [N=606,231] | 15 | 4
  T-BIL, PRE Below [N=606,231] | 0 | 0
  T-BIL, PRE Normal [N=606,231] | 587 | 224
  T-BIL, PRE Above [N=606,231] | 4 | 3
  T-BIL, Day 42 Unknown [N=583,220] | 16 | 4
  T-BIL, Day 42 Below [N=583,220] | 0 | 0
  T-BIL, Day 42 Normal [N=583,220] | 558 | 214
  T-BIL, Day 42 Above [N=583,220] | 9 | 2
  T-BIL, Day 182 Unknown [N=304,110] | 6 | 0
  T-BIL, Day 182 Below [N=304,110] | 0 | 0
  T-BIL, Day 182 Normal [N=304,110] | 296 | 110
  T-BIL, Day 182 Above [N=304,110] | 2 | 0
  T-BIL, Day 385 Unknown [N=251,104] | 7 | 1
  T-BIL, Day 385 Below [N=251,104] | 0 | 0
  T-BIL, Day 385 Normal [N=251,104] | 240 | 102
  T-BIL, Day 385 Above [N=251,104] | 4 | 1
  BIL-C/D, PRE Unknown [N=606,231] | 15 | 4
  BIL-C/D, PRE Below [N=606,231] | 0 | 0
  BIL-C/D, PRE Normal [N=606,231] | 591 | 226
  BIL-C/D, PRE Above [N=606,231] | 0 | 1
  BIL-C/D, Day 42 Unknown [N=583,220] | 16 | 4
  BIL-C/D, Day 42 Below [N=583,220] | 0 | 0
  BIL-C/D, Day 42 Normal [N=583,220] | 558 | 214
  BIL-C/D, Day 42 Above [N=583,220] | 9 | 2
  BIL-C/D, Day 182 Unknown [N=304,110] | 7 | 0
  BIL-C/D, Day 182 Below [N=304,110] | 0 | 0
  BIL-C/D, Day 182 Normal [N=304,110] | 297 | 110
  BIL-C/D, Day 182 Above [N=304,110] | 0 | 0
  BIL-C/D, Day 385 Unknown [N=251,104] | 8 | 1
  BIL-C/D, Day 385 Below [N=251,104] | 0 | 0
  BIL-C/D, Day 385 Normal [N=251,104] | 240 | 103
  BIL-C/D, Day 385 Above [N=251,104] | 3 | 0

32. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical Parameters Assessed With Respect to Creatinine (CREA) and Blood Urea Nitrogen (BUN)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  CREA, PRE Unknown [N=606,231] | 15 | 4
  CREA, PRE Below [N=606, 231] | 142 | 61
  CREA, PRE Within [N=606, 231] | 447 | 165
  CREA, PRE Above [N=606, 231] | 2 | 1
  CREA, Day 42 Unknown [N=583,220] | 17 | 4
  CREA, Day 42 Below [N=583,220] | 130 | 48
  CREA, Day 42 Within [N=583,220] | 432 | 166
  CREA, Day 42 Above [N=583,220] | 4 | 2
  CREA, Day 182 Unknown [N=304,110] | 6 | 1
  CREA, Day 182 Below [N=304,110] | 66 | 26
  CREA, Day 182 Within [N=304,110] | 231 | 83
  CREA, Day 182 Above [N=304,110] | 1 | 0
  CREA, Day 385 Unknown [N=251,104] | 6 | 0
  CREA, Day 385 Below [N=251,104] | 51 | 24
  CREA, Day 385 Within [N=251,104] | 191 | 80
  CREA, Day 385 Above [N=251,104] | 3 | 0
  BUN, PRE Unknown [N=606,231] | 15 | 4
  BUN, PRE Below [N=606,231] | 13 | 4
  BUN, PRE Within [N=606,231] | 553 | 218
  BUN, PRE Above [N=606,231] | 25 | 5
  BUN, Day 42 Unknown [N=583,220] | 17 | 4
  BUN, Day 42 Below [N=583,220] | 11 | 3
  BUN, Day 42 Within [N=583,220] | 531 | 209
  BUN, Day 42 Above [N=583,220] | 24 | 4
  BUN, Day 182 Unknown [N=304,110] | 6 | 0
  BUN, Day 182 Below [N=304,110] | 8 | 2
  BUN, Day 182 Within [N=304,110] | 281 | 105
  BUN, Day 182 Above [N=304,110] | 9 | 3
  BUN, Day 385 Unknown [N=251,104] | 7 | 0
  BUN, Day 385 Below [N=251,104] | 3 | 2
  BUN, Day 385 Within [N=251,104] | 237 | 100
  BUN, Day 385 Above [N=251,104] | 4 | 2

33. Secondary Outcome: Number of Subjects With Normal and Abnormal Haematological Parameters Assessed With Respect to Basophils (BAS) and Eosinophils (EOS)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  BAS, PRE Unknown [N=606,231] | 29 | 12
  BAS, PRE Below [N=606,231] | 0 | 0
  BAS, PRE Within [N=606,231] | 576 | 219
  BAS, PRE Above [N=606,231] | 1 | 0
  BAS, Day 42 Unknown [N=583,220] | 34 | 13
  BAS, Day 42 Below [N=583,220] | 0 | 0
  BAS, Day 42 Within [N=583,220] | 549 | 207
  BAS, Day 42 Above [N=583,220] | 0 | 0
  BAS, Day 182 Unknown [N=304,110] | 17 | 2
  BAS, Day 182 Below [N=304,110] | 0 | 0
  BAS, Day 182 Within [N=304,110] | 287 | 108
  BAS, Day 182 Above [N=304,110] | 0 | 0
  BAS, Day 385 Unknown [N=251,104] | 6 | 3
  BAS, Day 385 Below [N=251,104] | 0 | 0
  BAS, Day 385 Within [N=251,104] | 245 | 101
  BAS, Day 385 Above [N=251,104] | 0 | 0
  EOS, PRE Unknown [N=606,231] | 29 | 12
  EOS, PRE Below [N=606,231] | 68 | 19
  EOS, PRE Within [N=606,231] | 473 | 187
  EOS, PRE Above [N=606,231] | 36 | 13
  EOS, Day 42 Unknown [N=583,220] | 34 | 13
  EOS, Day 42 Below [N=583,220] | 49 | 15
  EOS, Day 42 Within [N=583,220] | 452 | 175
  EOS, Day 42 Above [N=583,220] | 48 | 17
  EOS, Day 182 Unknown [N=304,110] | 17 | 2
  EOS, Day 182 Below [N=304,110] | 33 | 11
  EOS, Day 182 Within [N=304,110] | 237 | 85
  EOS, Day 182 Above [N=304,110] | 17 | 12
  EOS, Day 385 Unknown [N=251,104] | 6 | 3
  EOS, Day 385 Below [N=251,104] | 32 | 17
  EOS, Day 385 Within [N=251,104] | 198 | 77
  EOS, Day 385 Above [N=251,104] | 15 | 7

34. Secondary Outcome: Number of Subjects With Normal and Abnormal Haematological Parameters Assessed With Respect to Haematocrit (Hcr) and Haemoglobin (Hgb)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  Hcr, PRE Unknown [N=606,231] | 26 | 10
  Hcr, PRE Below [N=606,231] | 53 | 21
  Hcr, PRE Within [N=606,231] | 480 | 181
  Hcr, PRE Above [N=606,231] | 47 | 19
  Hcr, Day 42 Unknown [N=583,220] | 19 | 7
  Hcr, Day 42 Below [N=583,220] | 45 | 13
  Hcr, Day 42 Within [N=583,220] | 477 | 178
  Hcr, Day 42 Above [N=583,220] | 42 | 22
  Hcr, Day 182 Unknown [N=304,110] | 12 | 2
  Hcr, Day 182 Below [N=304,110] | 38 | 7
  Hcr, Day 182 Within [N=304,110] | 238 | 91
  Hcr, Day 182 Above [N=304,110] | 16 | 10
  Hcr, Day 385 Unknown [N=251,104] | 5 | 3
  Hcr, Day 385 Below [N=251,104] | 18 | 12
  Hcr, Day 385 Within [N=251,104] | 215 | 85
  Hcr, Day 385 Above [N=251,104] | 13 | 4
  Hgb, PRE Unknown [N=606,231] | 26 | 10
  Hgb, PRE Below [N=606,231] | 61 | 26
  Hgb, PRE Within [N=606,231] | 497 | 182
  Hgb, PRE Above [N=606,231] | 22 | 13
  Hgb, Day 42 Unknown [N=583,220] | 19 | 8
  Hgb, Day 42 Below [N=583,220] | 69 | 19
  Hgb, Day 42 Within [N=583,220] | 476 | 185
  Hgb, Day 42 Above [N=583,220] | 19 | 8
  Hgb, Day 182 Unknown [N=304,110] | 11 | 2
  Hgb, Day 182 Below [N=304,110] | 42 | 16
  Hgb, Day 182 Within [N=304,110] | 241 | 89
  Hgb, Day 182 Above [N=304,110] | 10 | 3
  Hgb, Day 385 Unknown [N=251,104] | 5 | 3
  Hbg, Day 385 Below [N=251,104] | 27 | 15
  Hbg, Day 385 Within [N=251,104] | 210 | 84
  Hbg, Day 385 Above [N=251,104] | 9 | 2

35. Secondary Outcome: Number of Subjects With Normal and Abnormal Haematological Parameters Assessed With Respect to Neutrophils (NEU) and Platelets (PLA)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  NEU, PRE Unknown [N=606,231] | 29 | 12
  NEU, PRE Below [N=606,231] | 26 | 10
  NEU, PRE Within [N=606,231] | 534 | 202
  NEU, PRE Above [N=606,231] | 17 | 7
  NEU, Day 42 Unknown [N=583,220] | 34 | 13
  NEU, Day 42 Below [N=583,220] | 29 | 8
  NEU, Day 42 Within [N=583,220] | 505 | 189
  NEU, Day 42 Above [N=583,220] | 15 | 10
  NEU, Day 182 Unknown [N=304,110] | 17 | 2
  NEU, Day 182 Below [N=304,110] | 14 | 3
  NEU, Day 182 Within [N=304,110] | 266 | 105
  NEU, Day 182 Above [N=304,110] | 7 | 0
  NEU, Day 385 Unknown [N=251,104] | 6 | 3
  NEU, Day 385 Below [N=251,104] | 12 | 3
  NEU, Day 385 Within [N=251,104] | 227 | 96
  NEU, Day 385 Above [N=251,104] | 6 | 2
  PLA, PRE Unknown [N=606,231] | 35 | 17
  PLA, PRE Below [N=606,231] | 3 | 0
  PLA, PRE Within [N=606,231] | 518 | 187
  PLA, PRE Above [N=606,231] | 50 | 27
  PLA, Day 42 Unknown [N=583,220] | 32 | 12
  PLA, Day 42 Below [N=583,220] | 1 | 0
  PLA, Day 42 Within [N=583,220] | 500 | 184
  PLA, Day 42 Above [N=583,220] | 50 | 24
  PLA, Day 182 Unknown [N=304,110] | 20 | 5
  PLA, Day 182 Below [N=304,110] | 0 | 0
  PLA, Day 182 Within [N=304,110] | 260 | 96
  PLA, Day 182 Above [N=304,110] | 24 | 9
  PLA, Day 385 Unknown [N=251,104] | 8 | 8
  PLA, Day 385 Below [N=251,104] | 1 | 0
  PLA, Day 385 Within [N=251,104] | 234 | 94
  PLA, Day 385 Above [N=251,104] | 8 | 2

36. Secondary Outcome: Number of Subjects With Normal and Abnormal Haematological Parameters Assessed With Respect to Lymphocytes (LYM) and Monocytes (MON)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  LYM, PRE Unknown [N=606,231] | 29 | 12
  LYM, PRE Below [N=606,231] | 7 | 1
  LYM, PRE Within [N=606,231] | 441 | 161
  LYM, PRE Above [N=606,231] | 129 | 57
  LYM, Day 42 Unknown [N=583,220] | 34 | 13
  LYM, Day 42 Below [N=583,220] | 6 | 2
  LYM, Day 42 Within [N=583,220] | 446 | 162
  LYM, Day 42 Above [N=583,220] | 97 | 43
  LYM, Day 182 Unknown [N=304,110] | 17 | 2
  LYM, Day 182 Below [N=304,110] | 0 | 1
  LYM, Day 182 Within [N=304,110] | 235 | 93
  LYM, Day 182 Above [N=304,110] | 52 | 14
  LYM, Day 385 Unknown [N=251,104] | 6 | 3
  LYM, Day 385 Below [N=251,104] | 0 | 0
  LYM, Day 385 Within [N=251,104] | 223 | 86
  LYM, Day 385 Above [N=251,104] | 22 | 15
  MON, PRE Unknown [N=606,231] | 29 | 12
  MON, PRE Below [N=606,231] | 94 | 46
  MON, PRE Within [N=606,231] | 480 | 170
  MON, PRE Above [N=606,231] | 3 | 3
  MON, Day 42 Unknown [N=583,220] | 34 | 13
  MON, Day 42 Below [N=583,220] | 110 | 37
  MON, Day 42 Within [N=583,220] | 434 | 167
  MON, Day 42 Above [N=583,220] | 5 | 3
  MON, Day 182 Unknown [N=304,110] | 17 | 2
  MON, Day 182 Below [N=304,110] | 61 | 20
  MON, Day 182 Within [N=304,110] | 221 | 88
  MON, Day 182 Above [N=304,110] | 5 | 0
  MON, Day 385 Unknown [N=251,104] | 6 | 3
  MON, Day 385 Below [N=251,104] | 31 | 18
  MON, Day 385 Within [N=251,104] | 211 | 83
  MON, Day 385 Above [N=251,104] | 3 | 0

37. Secondary Outcome: Number of Subjects With Normal and Abnormal Haematological Parameters Assessed With Respect to Red and White Blood Cells (RBC and WBC)
Description: as for outcome 30
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject
  RBC, PRE Unknown [N=606,231] | 26 | 10
  RBC, PRE Below [N=606,231] | 25 | 4
  RBC, PRE Within [N=606,231] | 504 | 198
  RBC, PRE Above [N=606,231] | 51 | 19
  RBC, Day 42 Unknown [N=583,220] | 19 | 8
  RBC, Day 42 Below [N=583,220] | 21 | 6
  RBC, Day 42 Within [N=583,220] | 496 | 189
  RBC, Day 42 Above [N=583,220] | 47 | 17
  RBC, Day 182 Unknown [N=304,110] | 11 | 2
  RBC, Day 182 Below [N=304,110] | 13 | 5
  RBC, Day 182 Within [N=304,110] | 266 | 93
  RBC, Day 182 Above [N=304,110] | 14 | 10
  RBC, Day 385 Unknown [N=251,104] | 5 | 3
  RBC, Day 385 Below [N=251,104] | 8 | 2
  RBC, Day 385 Within [N=251,104] | 214 | 90
  RBC, Day 385 Above [N=251,104] | 24 | 9
  WBC, PRE Unknown [N=606,231] | 29 | 12
  WBC, PRE Below [N=606,231] | 27 | 9
  WBC, PRE Within [N=606,231] | 543 | 207
  WBC, PRE Above [N=606,231] | 7 | 3
  WBC, Day 42 Unknown [N=583,220] | 34 | 13
  WBC, Day 42 Below [N=583,220] | 38 | 8
  WBC, Day 42 Within [N=583,220] | 508 | 198
  WBC, Day 42 Above [N=583,220] | 3 | 1
  WBC, Day 182 Unknown [N=304,110] | 17 | 2
  WBC, Day 182 Below [N=304,110] | 21 | 7
  WBC, Day 182 Within [N=304,110] | 264 | 101
  WBC, Day 182 Above [N=304,110] | 2 | 0
  WBC, Day 385 Unknown [N=251,104] | 6 | 3
  WBC, Day 385 Below [N=251,104] | 15 | 6
  WBC, Day 385 Within [N=251,104] | 230 | 94
  WBC, Day 385 Above [N=251,104] | 0 | 1

38. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. "Any" was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period following Dose 1 of vaccine/placebo
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject | 153 | 63

39. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: as for outcome 38
Time Frame: During the 21-day (Days 21-41) post-vaccination period following Dose 2 of vaccine/placebo
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Influenza A (H5N1) Adjuvanted Group: This group results from the pooling of the Influenza A (H5N1) adjuvanted 6-<36M, Influenza A (H5N1) adjuvanted 3-<9Y and PInfluenza A (H5N1) adjuvanted 9-<18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (< 12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (>=) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 593 | 224
Subject | 135 | 54

40. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: as for outcome 38
Time Frame: During the 42-day (Days 0-41) post-vaccination period following Dose 1 of vaccine/placebo
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject | 243 | 97

41. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: A SAE was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 up to Day 385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group
Number analyzed (Participants) | 607 | 231
Subject | 8 | 4

42. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: as for outcome 38
Time Frame: During the 21-day (Days U0-U20) post-vaccination period following Dose 1 of Influenza A (H5N1) Virus monovalent vaccine
Population: as for outcome 19
Measure: Number; unit: Subject
Groups:
- Placebo/Influenza A (H5N1) Virus Monovalent Vaccine Group: Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6-<36M, Placebo 3-<9Y or Placebo 9-<18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9-<18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
Arm/Group | Placebo/Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 155
Subject | 21

43. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: as for outcome 38
Time Frame: During the 21-day (Days U21-U41) post-vaccination period following Dose 2 of Influenza A (H5N1) Virus monovalent vaccine
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Placebo/Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 155
Subject | 27

44. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. "Any" was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. As the study is still ongoing and data per age group are not available, results are presented for the groups pooled by vaccine/placebo administered. This outcome measure will be amended when data by age group become available.
Time Frame: During the 42-day (Days U0-U41) post-vaccination period following Dose 1 of Influenza A (H5N1) Virus monovalent vaccine
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Placebo/Influenza A (H5N1) Virus Monovalent Vaccine Group
Number analyzed (Participants) | 155
Subject | 41

45. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 41
Time Frame: From Day U0 up to Day U385
Population: as for outcome 19
Measure: Number; unit: Subject
Arm/Group | Placebo/Influenza A (H5N1) Adjuvanted Group
Number analyzed (Participants) | 155
Subject | 2

ADVERSE EVENTS:
Time Frame: Serious Adverse events (SAE) = Day 0 to Day 385 and Day U0 to U385. Solicited local and general symptoms = During the 7-day period post vaccine/placebo administration. Unsolicited AEs = During the 42-day post vaccine/placebo administration.
Description: For the systematically assessed other (non-serious) adverse events, number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Groups:
- Influenza A (H5N1) Adjuvanted Group: This group results from the pooling of the Influenza A (H5N1) adjuvanted 6-<36M, Influenza A (H5N1) adjuvanted 3≤9Y and Influenza A (H5N1) adjuvanted 9≤18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A vaccine or GSK Biologicals' monovalent A/Indonesia/5/2005 (H5N1) vaccine adjuvanted) at Days 0 and 21. Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. For children aged up to 12 months, 12 months excluded (<12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (≥12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
- Placebo Group: This group results from the pooling of the Placebo 6-<36M, Placebo 3-<9Y and Placebo 9≤18Y groups and includes subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who received 2 doses of 2 doses of saline placebo at Days 0 and 21. The saline placebo was administered intramuscularly. For children aged up to 12 months, 12 months excluded (<12 months), Dose 1 was administered in the left anterolateral thigh and Dose 2 in the right anterolateral thigh. For children older than (≥) 12 months, Dose 1 was administered in the deltoid region of the non-dominant arm (or left arm if dominance was not yet identified) and Dose 2 in the deltoid region of the dominant arm (or right arm).
- Placebo/Influenza A (H5N1) Adjuvanted Group: Subjects in this group were those who were administered the saline placebo solution in the Blinded Phase of the study (either in the Placebo 6≤36M, Placebo 3≤9Y or Placebo 9≤18Y Group). These were subjects aged at enrolment between 6 months and 18 years, 18 years excluded, who had received 2 doses of saline placebo at Days 0 and 21 in the Blinded Phase of the study, as per described in the descriptions of the Placebo 6≤36M, Placebo 3≤9Y and Placebo 9≤18Y groups. After consenting to participating to the Unblinded Phase of the study, these subjects received in addition 2 doses of Influenza A (H5N1) Virus monovalent vaccine at Days 385 (Day U0) and Day 385 + 21 days (Day U21). Influenza A (H5N1) Virus monovalent vaccine was administered intramuscularly. Dose 1 was administered in the deltoid region of the non-dominant arm and Dose 2 in the deltoid region of the dominant arm.
Arm/Group | Influenza A (H5N1) Adjuvanted Group | Placebo Group | Placebo/Influenza A (H5N1) Adjuvanted Group
Serious Adverse Events (participants affected / at risk) | 8/607 | 4/231 | 2/155
Other Adverse Events (participants affected / at risk) | 502/607 | 189/231 | 124/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza A (H5N1) Adjuvanted Group (N=607) | Placebo Group (N=231) | Placebo/Influenza A (H5N1) Adjuvanted Group (N=155)
Infectious mononucleosis (Infections and infestations) | 2 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group..
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Influenza (Infections and infestations) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Pneumonia (Infections and infestations) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 (0) — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Scarlet fever (Infections and infestations) | 0 | 0 | 1 — SAE assesed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 — SAE assessed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U385 for the Placebo/Influenza A (H5N1) adjuvanted Group.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Influenza A (H5N1) Adjuvanted Group (N=607) | Placebo Group (N=231) | Placebo/Influenza A (H5N1) Adjuvanted Group (N=155)
Pain (General disorders) | 405/603 | 69/229 | 111/154 — AE assesed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Swelling (General disorders) | 41/603 | 1/229 | 5/154 — AE assesed during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Drowsiness (General disorders) | 101/294 | 29/122 | 23/79 — AE assesed in children less than 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Irritability/fussiness (General disorders) | 128/294 | 40/122 | 28/79 — AE assesed in children less than 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Loss of appetite (General disorders) | 79/294 | 29/122 | 18/79 — AE assesed in children less than 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Fever (axillary temperature >= 38.0°C) (General disorders) | 59/294 | 21/122 | 4/79 — AE assesed in children less than 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Fatigue (General disorders) | 89/309 | 19/107 | 18/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Gastrointestinal disorders (General disorders) | 43/309 | 18/107 | 7/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Headache (General disorders) | 100/309 | 18/107 | 24/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Joint pain at other location (General disorders) | 50/309 | 9/107 | 14/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Muscle aches (General disorders) | 123/309 | 17/107 | 34/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Shivering (General disorders) | 25/309 | 7/107 | 7/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Sweating (General disorders) | 25/309 | 4/107 | 5/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Fever (axillary temperature >= 38.0°C) (General disorders) | 19/309 | 3/107 | 1/75 — AE assesed in children at least 6 years of age during Day 0 to Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 17 | 9 — AE assesed within the 42-day post-vaccination period following the first vaccination during Day 0 - Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Nasopharyngitis (Infections and infestations) | 29 | 18 | 10 — AE assesed within the 42-day post-vaccination period following the first vaccination during Day 0 - Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 27 | 13 | 3 — AE assesed within the 42-day post-vaccination period following the first vaccination during Day 0 - Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.
Diarrhoea (Gastrointestinal disorders) | 13 | 12 | 3 — AE assesed within the 42-day post-vaccination period following the first vaccination during Day 0 - Day 385 for Influenza A (H5N1) adjuvanted and Placebo Groups and from Day U0 to U42 for the Placebo/Influenza A (H5N1) adjuvanted Group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.